CLINICAL TRIAL: NCT02399488
Title: Validation of a Continuous Noninvasive Haemoglobin Determination Monitor (Radical 7 Pulse CO-Oximeter, SpHb) Compared to the Central Laboratory Coulter (LabHb) and a Point of Care (POC) Invasive Cooximeter (COoxHb) After in Vivo Adjustment.
Brief Title: Validation of Continuous Noninvasive Haemoglobin Monitoring by the Radical 7 Pulse CO-Oximetry Monitor After in Vivo Adjustment.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Juan Soliveres, MD, PhD, Hospital Universitario Doctor Peset
Other Study IDs: CEIC:47/10
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Sphb Haemoglobin in Vivo Validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Masimo Radical 7 — Simultaneous determination of haemoglobin with the continuous haemoglobin monitor, the central lanboratory coulter and a POC:

SUMMARY:
Continuous haemoglobin determination could improve the outcomes of several patients in risk of bleeding during surgery. An in vivo calibration has been introduced to the device after our team found its need. The uncalilbrated validation of the Masimo Radical 7 continuous haemoglobin monitor has been made in various papers, although it has been compared to point of care devices, thus introducing an error as such point of care devices although validated for haemoglobin determination, are not as accurate as the gold standard. The validation of the gold standard calibrated device has not been described yet.

When compared to the accepted gold standard (cyanmethemoglobin method, Coulter), accuracy and precision of the continuous haemoglobin monitor could be good enough to be used interchangeably with the gold standard.

DETAILED DESCRIPTION:
Continuous haemoglobin determination could improve the outcomes of several patients in risk of bleeding during surgery.

The in vivo calibration has not been adjusted to the gold standard haemoglobin determination in the literature yet.

Two blood samples will be withdrawn at the same time from an arterial line, one for the central laboratory and the other one for the POC device. At the same exact time the SpHb measurement will be recorded. At least eight samples are expected per patient. A maximum of 20 samples will be withdrawn per patient.

To compare bias, precision and limits of agreement among SpHb, LabHb and COoxHb the Bland Altman method will be used with multiple observations per subject when the true value varies. An error grid analysis will be made to know how it could affect to clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Surgery duration of at least two hours.
* Patients scheduled to surgery under general anaesthesia and muscle relaxation.
* Radial arterial line needed for blood pressure control or other reason not related to the study.

Exclusion Criteria:

* Radial arterial line not indicated / not possible to place.
* Sampling difficult or impossible.
* Need to reposition arterial line arm during surgery.
* Any illness that could influence the haemoglobin measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to any surgery of at least three hours of duration.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Central coulter bias and limits of agreement | 3 months
  Bias and limits of agreement of SpHb compared to the central laboratory coulter
Central coulter bias and limits of agreement after in vivo calibration | 3 months
  Bias and limits of agreement of SpHb compared to the central laboratory coulter after in vivo Radical 7 calibration

SECONDARY OUTCOMES:
POC Cooximeter bias and limits of agreement | 3 months
  Bias and limits of agreement of SpHb compared to the POC cooximeter
POC Cooximeter bias and limits of agreement | 3 months
  Bias and limits of agreement compared to the POC cooximeter after in vivo Radical 7 calibration
POC Cooximeter Coulter interchangeability | 3 months
  Bias and limits of agreement of POC Cooximeter Hb determination compared to the central laboratory coulter

OTHER OUTCOMES:
Comparison of bias and limits of agreement | 3 months
  Comparison of bias and limits of agreement among central laboratory, POC cooximeter and SpHb continuous monitor.
Clinical decision making | 3 months
  Error grid analysis plot

CONTACTS AND LOCATIONS:
Overall Officials: Juan Soliveres, MD, PhD, Principal Investigator — University Hospital Doctor Peset
Locations (1):
- University Hospital Doctor Peset, Valencia, Spain

REFERENCES:
- [Background] Soliveres J, Balaguer J, Estruch M, Sánchez A, Sánchez J. Validation of Continuous and Noninvasive Hemoglobin Monitoring from Pulse CO-Oximetry during Surgery. 2010 Annual Meeting of the American Society Anesthesiologists
- See also: Citation link — http://www.asaabstracts.com/strands/asaabstracts/searchArticle.htm;jsessionid=98A190E84BD2C1C22ECFC84E616E28D4?index=0&highlight=true&highlightcolor=0&bold=true&italic=false